CLINICAL TRIAL: NCT07091240
Title: Innovative Risk Calculator and Telehealth Delivered Parenting Program for Mental Health Promotion in Pediatric Primary Care: A Hybrid Type 3 Effectiveness-Implementation Study
Brief Title: Pediatricians Building Resilience Through Early Identification for Toddler Well-Being
Acronym: Peds-BRITE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Justin D. Smith, Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P50MH122402-PB; P50MH132502 (NIH)
Record Dates: First submitted 2025-07-09; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Check-up Online (FCU-O) (Experimental): In this study, caregivers of toddlers with a high likelihood of developing mental health challenges will participate in a parenting program, Family Check-Up® Online (FCU-O), and complete assessments related to their child's behavior and their caregiving practices. FCU-O is a parenting support program that offers tools and guidance to support children's emotional and behavioral development. The program is delivered through a secure website that can be accessed via computer or phone at participating caregivers' convenience. Caregivers will complete the Developmental Early Childhood Instrument for Deciding Effectively about Mental Health (DECIDE) tool, a risk calculator that screens for early signs of future mental health challenges, at their child's 24- or 30-month well-check visit with their pediatrician. Clinicians will use the DECIDE tool risk calculator score to refer caregivers of at-risk children to FCU-O. Caregivers may use FCU-O independently, or they may work with a trained coa
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Family Check-Up® Online is delivered through a secure website that can be accessed via computer or phone at participating caregivers' convenience. Caregivers will complete the Developmental Early Childhood Instrument for Deciding Effectively about Mental Health (DECIDE) tool, a risk calculator that screens for early signs of future mental health challenges, at their child's 24- or 30-month well-check visit with their pediatrician. Clinicians will use the DECIDE tool risk calculator score to refer caregivers of at-risk children to FCU-O. Caregivers may use FCU-O independently, or they may work with a trained coach who will facilitate their use of the program. Participation is open to caregivers who are referred to FCU-O based on their DECIDE risk calculator score by their child's pediatrician and is available in English or Spanish. Participants will also complete assessments via survey and direct observation before beginning FCU-O, and 6- and 12-months after their referral to FCU-O.

SUMMARY:
In this study, caregivers of toddlers with a high likelihood of developing mental health challenges will participate in a parenting program, Family Check-Up® Online (FCU-O), and complete assessments related to their child's behavior and their caregiving practices. FCU-O is a parenting support program that offers tools and guidance to support children's emotional and behavioral development. The program is delivered through a secure website that can be accessed via computer or phone at participating caregivers' convenience. Caregivers will complete the Developmental Early Childhood Instrument for Deciding Effectively about Mental Health (DECIDE) tool, a risk calculator that screens for early signs of future mental health challenges, at their child's 24- or 30-month well-check visit with their pediatrician. Clinicians will use the DECIDE tool risk calculator score to refer caregivers of at-risk children to FCU-O. Caregivers may use FCU-O independently, or they may work with a trained coach who will facilitate their use of the program. Participation is open to caregivers who are referred to FCU-O based on their DECIDE risk calculator score by their child's pediatrician, and is available in English or Spanish. Participants will also complete assessments via survey and direct observation before beginning FCU-O, and 6- and 12-months after their referral to FCU-O.

ELIGIBILITY:
Inclusion Criteria:

* Parents of toddler ages 22 month to 39 months who screen elevate on the Developmental Early Childhood Instrument for Deciding Effectively about Mental Health (DECIDE) tool risk calculator in a participating health center's pediatric practice

Exclusion Criteria:

* Unable to complete measures and consent process in English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychiatric Symptoms and Diagnosis | 12 month
  Parent interview to assess psychiatric disorders in preschool age children also known as the PAPA.

SECONDARY OUTCOMES:
Early Regulation and Context Assessment (ERICA) | Baseline, 6- and 12 month
  ERICA stands for early regulation and context assessment which is a direct assessment of child regulation skills.
Multidimensional Assessments Profile Scale (Temper Loss) (MAPS-TL) | 12-month
  This is a survey of child temper loss and irritability. Parents report on children's behavior on a scale of children's irritable behaviors on a scale from zero (never) to five (many times each day). They also report on the impact of child irritability on a scale from zero (no problems) to three (severe problems). Scores are summed and higher scores indicate more irritability behaviors.
Strengths and Difficulties Questionnaire (SDQ) | Baseline, 6- and 12-month
  The SDQ is a brief child behavior screening questionnaire. Parents report on children's strengths and difficulties on a three point scale (not true, somewhat true and certainly true). They also report on the impact of these strengths and difficulties on a four point scale which varies (e.g., no/yes with minor difficulties, definite difficulties/severe difficulties; not at all, only a little, a medium amount, a great deal). The total difficulties score is on a scale of 0 to 40 with higher scores indicating more difficulties. Then the internalizing and externalizing scores range from zero to twenty with higher scores indicating more emotional and peer difficulties. The impact score ranges from zero to 10 with higher scores indicating greater impact on daily life.
Early Childhood Irritability Related Impairment (E-CRI) | 12-month
  Early Childhood Irritability Related Impairment parent interview of childhood irritability and tantrums.
Early Childhood-Patient-Reported Outcomes Measurement Information System- Effortful Control (EC-PROMIS-EF) | 6- and 12-month
  Parent reported measure of children's effortful control. There are six parent report items on child's frustration tolerance and flexibility each item is on a five point scale from never (meaning no frustration tolerance and flexibility) to always (e.g., always flexible).
Family Assets Survey | Baseline, 6-, 12 month
  Family assets questionnaire is filled in by parents. This questionnaire has three domains with questions pertaining to parenting young children, the child parent relationship and family traditions with items scored with a minimum value of 1 and maximum value of 5. Mean scores are calculated with higher scores on this survey are associated with "more assets/strengths" as it relates to supporting the child's early mental health.
Minnesota Executive Function Scale (MEFS) | Baseline, 6- and 12-months
  Direct assessment of executive functioning that is completed by children on an internet browser i.e., children complete a card sorting task.
Multidimensional assessment profiles- Early Assessment Screening for Irritability (MAPS-EASI) | Baseline and 6-month
  The MAPS-EASI is a shortened version MAPS-TL designed for clinical screening. Parents report on children's irritable behaviors on a scale of zero (never) to five (many times each day). They also report on the impact of irritability on a scale from zero (no problems) to three (severe problems). Scores are summed and higher scores indicate more irritability behaviors. There is a maximum score of 15 for irritable behaviors and there is a maximum score of 6 on impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes